CLINICAL TRIAL: NCT05944978
Title: Phase Ib/II Clinical Study of GNC-035 Tetra-specific Antibody Injection in Relapsed or Refractory Chronic Lymphocytic Leukemia and Other Hematological Malignancies
Brief Title: A Study of GNC-035 in Relapsed or Refractory Chronic Lymphocytic Leukemia and Other Hematological Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNC-035-105
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Chronic Lymphocytic Leukemia
Keywords: Hematological malignancies
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants receive GNC-035 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: GNC-035

INTERVENTIONS:
Drug: GNC-035 — GNC-035 was intravenously infused 2h to 4h, once a week (IV, QW), and a 3-week cycle was used.

SUMMARY:
An open-label, multicenter, phase Ib/II clinical trial was conducted to evaluate the safety, tolerability, pharmacokinetics/pharmacodynamics, and antitumor activity of GNC-035 quad-specific antibody injection in patients with relapsed or refractory chronic lymphocytic leukemia and other hematological malignancies

DETAILED DESCRIPTION:
Phase Ib: To observe the safety and tolerability of GNC-035 in patients with hematologic malignancies such as relapsed/refractory chronic lymphocytic leukemia, and to determine the dose-limiting toxicity (DLT) and maximum tolerated dose (MTD), or maximum dose if MTD is not reached (MAD), of GNC-035. To determine the recommended phase II dose (RP2D) in hematologic malignancies such as chronic lymphocytic leukemia. Phase II: To explore the efficacy of GNC-035 in patients with relapsed/refractory chronic lymphocytic leukemia and other hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can understand the informed consent form, voluntarily participate in and sign the informed consent form;
2. No gender limit;
3. Age: ≥18 years old (≤75 years old for climbing);
4. expected survival time ≥3 months;
5. Patients with hematological malignancies such as relapsed/refractory chronic lymphocytic leukemia confirmed by histology or cytology;
6. For relapsed or refractory chronic lymphocytic leukemia (CLL/SLL), specifically:

   Patients who have relapsed after at least one line of standard therapy or have no response to or intolerance to standard regimens; Patients with relapsed or refractory chronic lymphocytic leukemia who were not or were ineligible for/intolerant of other therapies according to investigator assessment.

   Relapsed and refractory were defined as follows:

   Relapse was defined as disease progression after a response to adequate treatment, including at least one regimen containing a BTK inhibitor.

   Refractory was defined as refractory to BTK inhibitor, failure to achieve remission after adequate treatment with BTK inhibitor-containing regimens (combination therapy or monotherapy), or disease progression during treatment or within 6 months after completion of adequate treatment.
7. For other patients with relapsed refractory non-Hodgkin lymphoma. These include:

   Patients who experience failure of at least two lines of therapy; Relapsed or refractory patients who are not or are ineligible for/intolerant of other therapies as judged by the investigator.

   Relapsed and refractory were defined as follows:

   Relapse was defined as disease progression after a response to adequate treatment, including at least one anti-CD20 monoclonal antibody.

   Refractory was defined as refractory to anti-CD20 monoclonal antibody, failure to achieve remission after adequate treatment with anti-CD20 monoclonal antibody (combination therapy or monotherapy), or disease progression during treatment or 6 months after completion of adequate treatment.

   Among them, "adequate treatment with anti-CD20 monoclonal antibody" refers to the completion of full cycle of anti-CD20 monoclonal antibody combined with chemotherapy according to pathological type and disease stage, or anti-CD20 monoclonal antibody monotherapy at a dose of 375 mg/m2 once a week for at least 4 injections. Progression during treatment required the completion of at least one cycle of anti-CD20 monoclonal antibody combined with chemotherapy or monotherapy if progression occurred during induction therapy. At least one dose was completed if progression occurred during maintenance therapy. "Response" included complete and partial responses.
8. CLL/SLL: peripheral blood leukemia cells ≥5.0×109/L; Or the long diameter of any lymph node lesion ≥1.5cm; Patients with non-Hodgkin's lymphoma had measurable disease at screening (nodal disease ≥1.5cm in the greatest dimension or extranodal disease > 1.0cm in the greatest dimension).
9. ECOG ≤2;
10. Toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0 (except alopecia);
11. Organ function within 7 days before the first dose:

    Bone marrow function (for patients with non-Hodgkin lymphoma only) : without blood transfusion, G-CSF (for 2 weeks), and medication correction within 7 days prior to screening; Absolute neutrophil count (ANC) ≥1.0×109/L (≥0.5×109/L if the subject has bone marrow infiltration); Hemoglobin ≥80 g/L (≥70g/L if the subject has bone marrow infiltration); Platelet count ≥75×109/L; Liver function: total bilirubin, ≤1.5 ULN (Gilbert's syndrome, ≤3 ULN), and aminotransferase (AST/ALT), ≤2.5 ULN (for those with liver tumor invasive changes, ≤5.0 ULN) without correction with hepatoprotective medication within 7 days before screening examination; Renal function: creatinine (Cr) ≤1.5 ULN or creatinine clearance (Ccr) ≥60 mL/ minute (based on center calculation criteria) Coagulation: activated partial thromboplastin time (APTT) ≤1.5×ULN Prothrombin time (PT) ≤1.5×ULN.
12. Female subjects of childbearing potential or male subjects with a fertile partner must use highly effective contraception from 7 days before the first dose until 12 weeks after the last dose. Female subjects of childbearing potential must have a negative serum/urine pregnancy test within 7 days before the first dose;
13. Participants were able and willing to comply with protocol-specified visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

1. Patients who underwent major surgery within 28 days before study administration or who were scheduled to undergo major surgery during the study (" major surgery "was defined by the investigator);
2. Pulmonary disease grade ≥3 according to NCI-CTCAE v5.0, including dyspnea at rest or requiring continuous oxygen therapy; Patients with current interstitial lung disease (ILD) (except those who have recovered from previous interstitial pneumonia);
3. Severe systemic infection occurred within 4 weeks before screening, including but not limited to severe pneumonia caused by fungi, bacteria, or viruses, bacteremia, or serious infectious complications;
4. Patients with active autoimmune disease or a history of autoimmune disease. Patients with type I diabetes mellitus, hypothyroidism that is stable with hormone-replacement therapy (including hypothyroidism due to autoimmune thyroid disease), psoriasis, or vitiligo that does not require systemic therapy, as deemed by the investigators, were excluded.
5. Patients with other malignant tumors within 3 years before the first drug administration, cured non-melanoma skin cancer in situ, superficial bladder cancer, cervical cancer in situ, gastrointestinal mucosal cancer, breast cancer, localized prostate cancer, and other patients without recurrence within 3 years were excluded.
6. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBsAg positive or HBcAb positive and HBV-DNA test ≥ central detection lower limit) or hepatitis C virus infection (HCV antibody positive and HCV-RNA≥ central detection lower limit);
7. Hypertension poorly controlled by medication (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
8. Left ventricular ejection fraction ≤45%, or history of major heart disease within 1 year:

   1. New York Heart Association (NYHA) class III or IV congestive heart failure;
   2. Acute coronary syndrome, myocardial infarction or bypass or stent surgery (except those judged by the investigator to be stable);
   3. Patients with unstable angina pectoris;
   4. QT prolongation (QTcf > 450 msec in men or > 470 msec in women), complete left bundle branch block, degree III atrioventricular block, and arrhythmia requiring medical intervention;
   5. Other cardiac conditions deemed by the investigator to be ineligible for enrollment.
9. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of GNC-035;
10. Women who are pregnant or breastfeeding;
11. Presence of central nervous system invasion;
12. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (ALLo-HSCT);
13. Autologous hematopoietic stem cell transplantation (Auto-HSCT) within 12 weeks before starting GNC-035 therapy;
14. Current use of immunosuppressive agents, including, but not limited to, cyclosporine, tacrolimus, etc., within 2 weeks or 5 half-life periods prior to GNC-035 treatment, whichever is shorter;
15. Received radiotherapy, macromolecular targeted drugs within 4 weeks before GNC-035 treatment; Chemotherapy and a small-molecule targeted agent were administered 2 weeks or within five half-lives before treatment, whichever was less.
16. Received anti-CD20 therapy within 4 weeks prior to GNC-035 therapy and is responding;
17. Received CAR-T therapy within 12 weeks before GNC-035 treatment;
18. Use of a study drug from another clinical trial within 4 weeks or 5 half-lives, whichever was shorter, before the trial dose;
19. Other circumstances that the investigator deemed inappropriate for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ib: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle .
Phase Ib: Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-035. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-035.
Phase Ib: Recommended Phase II Dose (RP2D) | Up to 21 days after the first dose
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of GNC-035.
Phase II: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of GNC-035 to the first date of either disease progression or death, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Phase Ib: Complete Response (CR) | Up to approximately 24 months
  Complete response (CR) is defined as all tumor target lesions disappeared, no new lesions appeared, and tumor markers were normal for at least 4 weeks.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of GNC-035. The type, frequency and severity of TEAE will be evaluated during the treatment of GNC-035.
Phase Ib: Cmax | Up to 21 days after the first dose
  Maximum Drug Concentration (Cmax) of GNC-035 will be investigated.
Phase Ib: Tmax | Up to 21 days after the first dose
  Time at Which the Maximum (Tmax) of GNC-035 will be investigated.
Phase Ib: AUC0-inf | Up to 21 days after the first dose
  Area Under the Curve（0-inf）of GNC-035 will be investigated.
Phase Ib: AUC0-T | Up to 21 days after the first dose
  Area Under the Curve（0-t）of GNC-035 will be investigated.
Phase Ib: CL | Up to 21 days after the first dose
  Rate of clearance of GNC-035 will be investigated.
Phase Ib: T1/2 | Up to 21 days after the first dose
  Half-life (T1/2) of GNC-035 will be investigated.
Phase Ib: Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-GNC-035 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, MS, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences; Shuhua Yi, PHD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China